CLINICAL TRIAL: NCT06919406
Title: Temporal Dynamics of Mindfulness Intervention for Emotional Distress: Daily Interventions and Assessments
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Associate Dean, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20250325
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Emotional Distress; Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MBIs Group (Experimental): provide standard audio instructions for mindfulness exercises, introduce the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge, and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression, and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for emotional distress(MIED）

INTERVENTIONS:
Behavioral: Mindfulness Intervention for emotional distress(MIED） — MIED is an eight-week program developed based on MBSR and the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders. MIED consists of weekly group sessions with daily interactive materials delivered via a WeChat-based mini-program. The group sessions, conducted online, provide structured content and interactive discussions aligned with the weekly themes, for example including psychoeducation on mindfulness, emotions, and emotional distress. Mini Program and lasted for 49 days. Each day, participants received different materials including (a) an audio recording of mindfulness meditation guidance; (b) learning materials in text or audio; and (c) assignments (for example, informal mindfulness practice, emotion journal, and challenging tasks).

SUMMARY:
This research aims to adopt a complex systems perspective to thoroughly examine the impact of online mindfulness interventions on changes in emotional distress, with a particular focus on the mechanisms of action. Through a daily diary study design, the study seeks to reveal the complexity and dynamic characteristics of emotional changes and the underlying mechanisms（i.e. distress tolerance， experiential avoidance， cognition flexibility, and life engagement） throughout the intervention process. This research will enrich the theoretical framework of online mental health intervention and provide empirical evidence for optimizing online intervention strategies.

DETAILED DESCRIPTION:
Emotional distress refers to psychological discomfort related to emotions-particularly anxiety and depression-as well as the associated suffering and impairments in work and daily life. According to a Gallup survey, approximately one-third of the global population experiences emotional distress (Daly & Macchia, 2023), with depression, anxiety, and anger being the most prominent aspects. Moreover, the distress associated with worry and sadness has increased significantly from 2009 to 2021. Anxiety disorders and depressive disorders are among the most common mental illnesses worldwide (Kessler et al., 2009; World Health Organization, 2017), and depression is the leading cause of suicide (Ferrari et al., 2014). In China, the lifetime prevalence rates for anxiety disorders and depression are approximately 7.5% and 6.8%, respectively (Y. Huang et al., 2019), with only about 0.5% of patients with depression receiving adequate treatment (Lu et al., 2021). Both anxiety and depressive disorders severely restrict psychosocial functioning and adversely affect normal life. Traditional psychotherapy research has largely been limited to phenomenological descriptions, lacking in-depth exploration of the underlying mechanisms, which in turn constrains the optimization and effectiveness of interventions.

The theories and methods from the field of complex systems can help overcome these limitations by providing a deeper theoretical framework and analytical tools for studying the processes and mechanisms underlying psychotherapeutic effects. In recent years, network analysis and dynamic systems research on psychological interventions for anxiety and depressive disorders have gradually advanced. However, most current studies collect data only before and after the intervention, paying little attention to the dynamic changes during the intervention period and the long-term impact during follow-up. At the network element level, most studies focus on symptom networks, with few incorporating mechanistic variables into their models. Understanding the mechanisms of intervention effects is critical, and this requires including more mechanistic variables in the analysis framework. In conjunction with dynamic systems theory, it is possible to further explore state transitions and their early warning signals. Although early warning signals theoretically hold the potential to predict sudden changes, their practical sensitivity and specificity still need to be improved in order to provide more reliable information for clinical practice.

In summary, existing research suggests that complex network methods hold potential value in clinical practice, warranting further exploration. However, current findings are insufficient to fully and deeply reveal the specific processes underlying psychotherapeutic effects (Holmes et al., 2018). Moreover, the practical utility of complex network methods in clinical settings remains to be verified (Contreras et al., 2019; Schreuder et al., 2023). This is particularly true in the field of mindfulness interventions, where research in this area is still lacking. By adopting a complex systems perspective, incorporating intensive longitudinal measurements, and including mechanistic variables（i.e. distress tolerance， experiential avoidance， cognition flexibility, and life engagement）, this study aims to explore feedback loops with temporal dynamic characteristics. Such an approach will enable researchers to gain a more comprehensive and in-depth understanding of the complexity and dynamics involved in the alleviation of emotional distress such as anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.

Exclusion Criteria:

* Subjects who could not access the Internet.
* Subjects with insufficient Chinese ability.
* Subjects who have participated in mindfulness-based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week.
* Patients with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder.
* Subjects at risk of suicide.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-05 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Daily changes of depression | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily Depression Severity and Impairment Scale,5 items, scores range from 0 to 20, with higher scores indicating higher levels of depression.
Daily changes of anxiety | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily Anxiety Severity and Impairment Scale,5 items, scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Daily changes of engaging in everyday life | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Self-developed scale assessing the extent to which individuals' daily engagement in life domains (such as work, social interactions, and leisure activities) is affected by physical and psychological discomfort, 4 items, scores range from 0 to 16, with higher scores indicating higher levels of engaging in everyday life.
Daily changes of distress tolerance | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Based on a preliminary study, the items with the highest factor loading from each subscale of the DTS (Simon & Gaher, 2005) were chosen to form the Daily Distress Tolerance Scale (DDTS). The DDTS consists of four items. Each item is rated on a scale ranging from 1 (strongly agree) to 5 (strongly disagree). Scores range from 4 to 20, with higher scores indicating greater distress tolerance.
Daily changes of cognitive flexibility | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Based on a preliminary study, the items with the highest factor loading from each subscale of the DTS (Dennis &Vander Wal，2010) were chosen to form the Daily Cognitive Flexibility Inventory (DCFI). The DCFI consists of 2 items，that is "I consider multiple options before making a decision"， "When I encounter difficult situations, I feel like I am losing control(reverse scored)". Each item is rated on a scale ranging from 1 (never) to 5 (always). After reverse scoring the second item, the scores are summed, resulting in a total score ranging from 2 to 10, with higher scores indicating greater cognitive flexibility.
Daily changes of treating thoughts as thoughts | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  self-developed questionnaire, measuring to what extent individuals could treat thoughts as psychological phenomena rather than facts, one item, scores range from 1 to 5, with higher scores indicating higher levels of treating thoughts as thoughts.
Daily changes of Experiential Avoidance | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Based on a preliminary study, the items with the high factor loading （at least higher than 0.6） from each subscale of the Brief Experiential Avoidance Questionnaire ( Gámez et al, 2013) were chosen to form the Daily Experiential Avoidance Scale (DEAS). The DEAS consists of four items. Each item is rated on a scale ranging from 1 (strongly agree) to 6 (strongly disagree). Scores range from 5 to 30, with higher scores indicating less experiential avoidance.
Daily changes of Emotion | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  Daily positive and negative affect were measured using the 10-item International Positive and Negative Affect Schedule-Short Form Scale. Scores range from 0 to 100, with higher scores indicating higher levels of positive/negative affect.
Daily changes of mindfulness | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  The Daily Mindfulness Response Scale measures the frequency with which one returns to a nonjudgmental and unconditionally receptive present moment awareness during the day. Each item is rated on a scale ranging from 1 (rarely) to 10 (often). scores range from 4 to 40, with higher scores indicating higher levels of mindful responding
Daily changes of repeative negative thinking | once per day for 63 days (1 week pre-intervention, 7 weeks during the intervention, 1 week post-intervention)
  4 items are adapted from the original Momentary Repetitive Negative Thinking Scale, rated on a scale from 1 (Not at all) to 8 (Very intensely). Total scores range from 4 to 32, where higher scores indicate greater severity of momentary repetitive negative thinking, reflecting more frequent and intense experiences of intrusive, uncontrollable negative thought cycles.

SECONDARY OUTCOMES:
changes of trait mindfulness | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
changes of Psychological Distress | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
changes of depression | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  The Patient Health Questionnaire-9 (PHQ-9) measures the severity of depressive symptoms over the past two weeks. Each item is rated on a scale ranging from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
changes of anxiety | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  The Generalized Anxiety Disorder-7 (GAD-7) measures the severity of generalized anxiety symptoms over the past two weeks. Each item is rated on a scale ranging from 0 (not at all) to 3 (nearly every day). Scores range from 0 to 21, with higher scores indicating greater severity of anxiety symptoms.
changes of Athens Insomnia Scale | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  The Athens Insomnia Scale is a self-reported questionnaire measuring sleepy quality. Scores range from 0 to 24, with lower scores indicating higher levels of sleep quality.
changes of engaging in everyday life | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  Self-developed scale assessing the extent to which individuals' daily engagement in life domains (such as work, social interactions, and leisure activities) is affected by physical and psychological discomfort. , 16 items, scores range from 0 to 64, with higher scores indicating higher levels of engaging in everyday life.
changes of Brief Experiential Avoidance Questionnaire | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  Chinese version of the Brief Experiential Avoidance Questionnaire scale is used to measure Experiential Avoidance.Scores range from 15 to 90, with higher scores indicating higher levels of experiential avoidance.
changes of Distress Tolerance Scale | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  Distress Tolerance Scale is used to measure Distress Tolerance. Scores range from 5 to 75, with higher scores indicating higher levels of Distress Tolerance.
changes of Overall Anxiety Severity and Impairment Scale | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
changes of Overall Depression Severity and Impairment Scale | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
changes of treating thoughts as thoughts | 1 week before the intervention, the onset of the intervention，1 week after the onset of the intervention，2 week after the onset of the intervention， 1 month after the intervention，3 month after the intervention
  The questionnaire has 1 dimension and contains 5 items on a five-point Likert scale (1=completely compliant, 5=completely non-compliant), with higher scores indicating higher ability to treat ideas as ideas.
changes of Cognitive flexibility Inventory | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  Cognitive flexibility Inventory is a self-reported questionnaire measuring Cognitive flexibility level.Scores range from 20 to 100, with higher scores indicating higher levels of Cognitive flexibility.
changes of Perseverative Thinking Questionnaire | 1 week before the intervention, 1 month after the intervention，3 month after the intervention
  Perseverative Thinking Questionnaire,16 items, scores range from 0 to 60, with higher scores indicating greater severity of repetitive negative thinking (RNT).

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University

IPD SHARING:
Plan to Share IPD: No